CLINICAL TRIAL: NCT02201277
Title: Prospective Randomized Evaluation of the Denali and Option Inferior Vena Cava Filters
Brief Title: ODEN Trial: Option vs. Denali IVC Filters
Acronym: ODEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ODEN trial stopped due to low enrollment & to focus on the PRESERVE Trial.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSF 14-13307
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Venous Thromboembolism
Keywords: IVC; IVC Filter; Filter; Option; Denali; filter tilt; filter migration; filter fracture; filter thrombus; filter penetration
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: analysis of the imaging data will be masked and filter type and PHI will be redacted so the radiologist assessor will not know which patients receive either the option or denali..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Denali (Experimental): Denali IVC Filter
  Interventions: Device: Filter Placed
- Option (Experimental): Option Elite IVC Filter
  Interventions: Device: Filter Placed

INTERVENTIONS:
Device: Filter Placed

SUMMARY:
This research study is a prospective randomized trial evaluating the relative safety of two inferior vena cava (IVC) filters used to prevent the migration of potentially dangerous deadly blood clots from the legs to the lung in patients who cannot take blood thinners. All eligible patients will have been ordered to have a IVC filter placed by their primary medical team and filters will be placed in these patients whether or not they wish to participate in this trial as part of standard of care. The investigators will follow up with patients 30 days after IVC filter placement and ask them to come back for filter removal if medically appropriate. If removal is not medically appropriate in 30 days, the investigators will attempt to schedule removal every 30 days after initial placement.

Primary outcome measures will be IVC filter complications such as filter penetration through the IVC wall and into other organs, filter tilt, filter migration, filter fracture and clots formed within the filter. All of these are reported complications of all IVC filters.

The research also aims to improve the standard of care for IVC filter patient follow up as the FDA and Society of Interventional Radiology recommend that IVC filters be removed as soon as it is safe to do so.

Hypothesis:

The investigators hypothesize that there is no significant difference in efficacy and complication rate between the Option and the Denali filter.

DETAILED DESCRIPTION:
This is a prospective, randomized trial comparing two FDA-approved inferior vena cava filters, the Denali retrievable IVC filter (Bard Peripheral Vascular Inc., Tempe, AZ) and the Option Elite (Argon Medical, Athens, Texas).

Patients scheduled for IVC filter placement at UCSF Department of Interventional Radiology (IR) will be asked by the IR physician performing the procedure at either UCSF Mt. Zion or Moffitt hospital if they wish to participate in this prospective, randomized study. Recruitment will be conducted by the physicians performing the IR procedures only. No additional recruitment calls, emails, posters or web pages are necessary. All procedures and the randomization to one of the two experimental groups will be carefully explained before obtaining signed written consent.

Screening:

Screening will be conducted by the IR physician prior to the placement of the IVC filters. Since this is a standard of care study, patients who are recommended for IVC filter placement and are scheduled for the procedure are generally eligible.

The screening procedures are part of routine care before IVC filter placement and would be done even if patients did not join the study.

The study doctor will review the results of most recent routine care imaging scans (CT or MRI) of the abdomen and pelvis. This is done to confirm that the diameter of IVC is no wider than 2.8cm. Both filters are FDA-approved to be placed in an IVC with maximal diameter of 2.8cm.

The study doctor will also review ultrasound of the lower extremity, when available, to confirm that a blood clot was in fact present prior to performing the study. This ensures that patients who present for IVC filter placement are screened properly.

The following screening procedures should be done within 12 days before the IVC filter placement procedure as part of the standard of care.

* A complete physical exam
* The study doctor will ask about medical history and how well patient is able to do daily activities
* Routine care blood tests (about 2 tablespoons) o This is to ensure that the INR and platelet count of the patient is within the safe limits to perform an invasive procedure.

After Enrollment:

If the screening procedures show that the patient is eligible and consents to take part in the study, IVC filter placement will occur after randomization.

After enrollment, the following procedures will be done during the study: Just as with screening, all of these procedures are part of regular IVC filter placement care.

Randomization:

Randomization will occur on the day of procedure or prior clinic visit with IR physician to either the Denali or Option IVC filter. All IR attending physicians on the protocol are familiar with placement of either filter type. Prior to opening study to accrual, 75 sealed security envelopes with the word Denali printed on a card inside and 75 sealed security envelopes with the word Option will be assembled by IR staff not involved in the research. The envelopes will be mixed up and placed in a bag. Computerized randomization programs and tables were considered but we feel the envelopes will work best as there may be limited time after patient is consented and procedure begins. This is especially true as some filters are placed emergently. Previous IR studies have used this randomization technique with great success.

Filter Placement:

Placement of an IVC filter involves the insertion of a plastic tube (catheter) into a vein in the neck. Some numbing medicine (Lidocaine) will be injected in the skin over the vein before the catheter is inserted. Intravenous medications will be given to induce moderate sedation (Fentanyl for analgesic and Versed for moderate sedation). Once the catheter has been placed into the vein, it will be advanced into the IVC. Once in correct position, x-ray contrast material (x-ray dye-Omnipaque 350) will be injected through the catheter and x-ray pictures taken. A series of x-ray pictures will be obtained of the IVC. These pictures are taken as part of standard of care to determine the position of the renal veins with respect to the IVC. The top of the filter must sit below the renal veins so it does not cause obstruction of the renal veins. In addition, pictures of the IVC are taken to serve as another tool in measuring the diameter of the IVC to make sure the diameter of the IVC is less than 2.8cm. This is particularly important in situations when a CT or MRI of the abdomen and pelvis is not available to have reviewed prior to the procedure. Once pictures are obtained and it is made certain that the IVC diameter is less than 2.8cm, the filter will be inserted through the catheter, and placed below the renal veins. During the placement procedure, positioning of the filter will be monitored with x-ray pictures. At the completion of the procedure the catheter will be removed and pressure will be applied to the insertion site until the bleeding has stopped. All of this is part of routine standard of care for placement of the filter. The doctor performing the procedure will be asked to complete a short questionnaire after IVC filter placement which will be attached to "Study Documents".

Follow-Up:

After the IVC filter placement procedure patient status will be followed by the interventional radiology doctors.

Per standard of care after IVC filter placement, patient will be monitored in the hospital for up to 1 hour after the procedure. If patient is in stable condition and sedation has resolved, they will return home the same day or returned to their hospital rooms.

A tentative appointment for follow up and filter retrieval will be ordered by IR physician at time of filter placement in APEX. This will ensure that scheduling and study staff will be aware that further patient and primary care follow-up is required.

Patient primary care physician and/or relevant medical staff will be telephoned one month after IVC filter placement to determine if patient is medically stable and suitable for IVC filter removal.

If IR and other doctors agree that IVC filter removal is recommended, patient will be scheduled to return for follow-up imaging and filter retrieval. If patient is not medically stable or still at high risk for blood clots, we will attempt to schedule a follow up one month later. Close contact with primary physician and patient will be maintained to ensure that filter is removed as soon as possible. APEX scheduling will be used to make sure follow up is performed at regular intervals.

At follow-up appointment these routine tests per standard of care before IVC filter removal will be performed:

* A physical exam
* The study doctor will ask about medical history, how well patient is able to do daily activities, and if they are experiencing any possible symptoms related to the IVC filter placement such as abdominal or back pain.
* A rotation CT focused to the site of the filter will be performed as part of routine practice of filter removal. This is done to ensure the filter has not migrated or that the filter has not penetrated through the walls of the IVC such that filter retrieval would be unsafe.
* IR physician will determine if patient status is stable and safe for IVC filter removal. If not, physician will discuss with primary care doctor if filter needs to remain permanently in patient or if later retrieval should be considered at subsequent follow up visits.
* IVC filter retrieval will be performed under moderate sedation. This procedure is very similar in nature to the filter placement procedure. The IVC filter is removed via a similar process to the way in which it was placed. X-ray dye (contrast) will be injected around the filter to assure that the filter and the area beneath the filter are free of blood clots and that it is safe to proceed with removal. A catheter-based snare will be used to engage the hook at the end of the filter and the filter will then be enveloped by a removal sheath and removed from the body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for IVC filter placement at UCSF Moffitt, Mission Bay and Mount Zion hospitals Interventional Radiology
2. 18+

Exclusion Criteria:

1. Necessity of permanent IVC filter.
2. Genetic or physical abnormalities of the inferior vena cava
3. Circumstances that in the opinion of the primary investigator, patient would be a poor candidate either due to complications in medical condition or lack of ability for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen P Kohi, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Woodcock A, Campbell I, Collins JV, Hanson P, Harvey J, Corris P, Johnston ID. Bronchoscopy and infection control. Lancet. 1989 Jul 29;2(8657):270-1. doi: 10.1016/s0140-6736(89)90451-0. No abstract available. PMID 2569071
- See also: ucsf radiology home page — http://radiology.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2014-May 2016, patients coming to University of California, San Francisco Interventional Radiology (IR) with a MD referral for an Inferior Vena Cava (IVC) filter were invited to join a study of two FDA approved filters. After informed consent, subjects were randomized 1:1 to receive either a Denali or Option Elite filter.
Units Other Than Participants: retrievable vena cava filters
Groups:
- Denali: Denali brand IVC Filter will be placed in patients randomized to Denali Arm.
- Option Elite: Option Elite brand IVC Filter will be placed in patients randomized to Option Arm.
Period: Overall Study
Arm/Group | Denali | Option Elite
Started | 24; 25 retrievable vena cava filters (24 patients were consented but 1 patient had denali filter placed twice.) | 21; 20 retrievable vena cava filters (1 patient was withdrawn after signing consent due to physician preference for the option filter.)
Filter Retrieval | 17; 17 retrievable vena cava filters | 16; 16 retrievable vena cava filters
Signed ICF But Did Not Enroll | 0; 0 retrievable vena cava filters (Physician had preference for a specific filter so patient not randomized.) | 1; 1 retrievable vena cava filters
Filter Ruled to be Permanent | 2; 2 retrievable vena cava filters | 2; 2 retrievable vena cava filters
Lost to Follow up | 2; 2 retrievable vena cava filters | 1; 1 retrievable vena cava filters
Death (Before Removal) (All cause mortality not related to the study devices.) | 3; 3 retrievable vena cava filters | 4; 4 retrievable vena cava filters
Complicated Retrieval (2 filters failed 1st attempts at retrieval then success.) | 2; 2 retrievable vena cava filters | 0; 0 retrievable vena cava filters
Failed Retrieval (Referred Elsewhere) | 1; 1 retrievable vena cava filters | 0; 0 retrievable vena cava filters
Completed | 17; 18 retrievable vena cava filters | 16; 16 retrievable vena cava filters
Not Completed | 7; 7 retrievable vena cava filters | 5; 4 retrievable vena cava filters
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Failed retrieval | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: 45 participants signed consent forms in the trial however one was withdrawn from the Option group due to physician's choice and in the Denali group one participant had two filters placed at different times.
Units Other Than Participants: filters
Groups:
- Option: Option Elite IVC Filter brand IVC Filter will be placed in patients randomized to Option Arm.
- Total: Total of all reporting groups
Arm/Group | Denali | Option | Total
Number analyzed (Participants) | 24 | 21 | 45
Number analyzed (filters) | 25 | 20 | 45
Age, Categorical [Count of Participants; unit: Participants] — age at enrollment
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 12 | 24
    >=65 years | 12 | 9 | 21
Sex: Female, Male [Count of Participants; unit: Participants] — *one male was not randomized
  Participants
    Female | 11 | 10 | 21
    Male | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 16 | 33
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45
Indication for filter placement [Count of Participants; unit: Participants] — In addition to known venous thromboembolism (VTE)
  Participants
    VTE and contraindication to anticoagulation | 13 | 11 | 24
    Prophylactic (no current thromboembolic disease) | 8 | 8 | 16
    Failure to maintain anti coagulation | 1 | 1 | 2
    Recurrent Pulmonary Embolism Despite Therapy | 1 | 1 | 2
    Complication from Anti coagulation | 1 | 0 | 1
Filter Indwelling Time [Mean (Full Range); unit: days since filter placement] | 378.7 [0 to 1647] | 277.1 [0 to 1733] | 331.3 [0 to 1733]

OUTCOME MEASURES:

1. Primary Outcome: IVC: Filter Penetration
Description: Using imaging analysis, patients will resume their standard care as normal but be encouraged to come back in 30 days for imaging followup and removal. other than that we will look at all available CT and xray imaging that clearly shows the filter and IVC vessel walls. We will count how many participants have penetration of the IVC greater than 3mm and the number of days since placement at imaging timepoints. The number of struts or hooks per filter with penetration will also be recorded.
Time Frame: in dwelling time in 1 day after filter insertion up to 3 years.
Population: patients consented to the trial and needing a temporary ivc filter
Measure: Number; unit: Participants
Groups:
- Denali: Denali filter randomized participants
- Option: Option filter randomized participants
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Participants | 24 | 20
Statistical Analysis 1: Comparison: Denali vs Option; A Fisher's exact test was used to determine if there was a difference in the numbers of filters with penetration for each type. The numbers were not powered enough to make extensive tests in this area meaningful; Test type: Superiority; p = 1.0, t-test, 2 sided
Statistical Analysis 2: Comparison: Denali vs Option; Test type: Equivalence — rate of penetration; p = 1.0, t-test, 1 sided

2. Secondary Outcome: Computerized Tomography (CT) Studies With IVC Penetration
Description: All CT studies with IVC penetration ≥ 3 mm, (%)
Time Frame: 0-1733 days
Population: Imaging was analyzed to see if filter penetration could be observed and there was some penetration on imaging but nothing beyond 3mm.
Measure: Number; unit: Penetrating filter struts
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Penetrating filter struts | 0 | 0

3. Secondary Outcome: Number of Participants With IVC Filter Migration
Description: The number of participants with IVC filter migration in terms of distance migrated from initial placement location 30 days after filter placement will be assessed radiographically.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Participants | 0 | 0

4. Secondary Outcome: IVC Filter Tilt
Description: number of participants with tilt of greater than 15 degrees in any CT imaging studies after filter placement and before removal of filter or study endpoint reached.
Time Frame: 0-365 days post placement until project closure or patient endpoint reached
Measure: Number; unit: participants
Groups:
- Denali Filter Tilt; Option Filter Tilt: # of participants with tilt greater than or equal to 15 degrees
Arm/Group | Denali Filter Tilt | Option Filter Tilt
Number analyzed (Participants) | 24 | 20
participants | 0 | 0

5. Secondary Outcome: IVC Filter Fracture
Description: Fracture of the component legs and struts of the IVC filter will be determined radiographically 30 days after placement.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Participants | 0 | 0

6. Secondary Outcome: IVC Filter Clot
Description: Thrombus (or clot) formed in the IVC filter 30 days after placement will be assessed radiographically.
Time Frame: 30 days
Population: the population sample size was not large enough to see differences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Participants | 2 | 2

7. Secondary Outcome: IVC Filter Improved Patient Follow Up and Prompt Filter Removal
Description: The research also aims to improve the standard of care for IVC filter patient follow up as the FDA and Society of Interventional Radiology (SIR) recommend that IVC filters be removed as soon as it is safe to do so. Ideally filters will be imaged and removed after 30 days but in some cases patients will need filters to remain in place longer. We will make every effort to encourage patients and their medical team to return for follow up imaging and filter removal as soon as is deemed medically safe.
Time Frame: Number of participants who had filters removed after 30 days up to 1 year
Measure: Number; unit: Filter
Units Other Than Participants: Filter
Groups:
- Denali: Denali IVC Filter
  Filters retrieved %
- Option: Option Elite IVC Filter
  Filter retrieved %
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Number analyzed (Filter) | 24 | 20
Filter | 17 | 16

8. Secondary Outcome: IVC Filter Improved Patient Follow Up and Prompt Filter Removal: Number of Days
Description: as for outcome 7
Time Frame: Number of participants who had filters removed after 30 days up to 1 year
Population: Participants
Measure: Number; unit: Days
Units Other Than Participants: Filter
Arm/Group | Denali | Option
Number analyzed (Participants) | 24 | 20
Number analyzed (Filter) | 24 | 20
Days | 161.7 | 130.8

ADVERSE EVENTS:
Time Frame: During the study, site personnel will note any change in the condition(s) and the occurrence and nature of any adverse events. For 30 days after removal of IVC filter or until study endpoint reached, patients will be followed for any adverse event that could be related to the IVC filter or removal.
Description: All adverse events (AE) attributed to the IVC filter device will be recorded until resolved or the AE is assessed as:
  * stable
  * new therapy started
  * patient lost to follow-up
  * withdraws
  * death
  All serious adverse events (SAE) related to trial-related procedures will be followed until a final outcome & resolution date is documented. If, after follow-up, return to baseline status or stabilization cannot be established before study exit an explanation should be recorded.
Groups:
- Denali: Denali brand IVC Filter will be placed in patients randomized to Denali Arm.
  24 enrolled
- Option: Option brand IVC Filter will be placed in patients randomized to Option Arm.
  22 enrolled 1 withdrawn by investigator after consent before randomization and 1 patient had 2 filters placed.
Arm/Group | Denali | Option
All-Cause Mortality (participants affected / at risk) | 4/24 | 3/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 0/24 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denali (N=24) | Option (N=20)
Filters with IVC penetration ≥ 3 mm (Vascular disorders) | 0 (0) | 0 (0) — # of filters placed with IVC penetration by hook or strut greater than or equal to 3mm
All CTs with IVC penetration (Vascular disorders) | 0 (0) | 0 (0) — # of CTs with IVC penetration greater than or equal to 3 mm.
Filter Fracture (Vascular disorders) | 0 (0) | 0 (0) — Filter fracture is any loss of a filter's structural integrity (ie, breakage or separation) documented by imaging or at autopsy
Filter movement (Vascular disorders) | 0 (0) | 0 (0) — Filter movement is a change in filter position compared with its deployed position (cranial or caudal) of more than 2 cm as documented by plain radiography, CT, or venography.
Filter Tilt > or = 15 deg. (Vascular disorders) | 0 (0) | 0 (0) — Patients with tilt greater than or equal to 15 degrees on greater than or equal to 1 CT study
All CT studies with Tilt (Vascular disorders) | 0 (0) | 0 (0) — All CT studies with tilted filters greater than or equal to 15 degrees

LIMITATIONS AND CAVEATS:
The ODEN trial was initially powered to observe differences between the two filter types after 75 of each filter were to be placed. Due to the opening of the PRESERVE trial and slightly lower than expected enrollment, the trial was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: IRB Application (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02201277/Prot_SAP_000.pdf
  • Informed Consent Form (2014-05-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02201277/ICF_001.pdf
  • Study Protocol: NCT02201277 References (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02201277/Prot_002.pdf